CLINICAL TRIAL: NCT00841932
Title: Retrospective Assessment of the Safety of Performing Fractional Flow Reserve (FFR) of the Myocardium Without Anticoagulation During Diagnostic Cardiac Catheterization
Brief Title: Performing Fractional Flow Reserve Without Anticoagulation During Diagnostic Catheterization
Status: Completed | Type: Observational
Sponsor: Clinyx, LLC (Other)
Collaborators: Volcano Corporation (Industry)
Responsible Party: Holly Taylor, VP, Clinyx
Other Study IDs: CL-002
Record Dates: First submitted 2009-02-06; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve; Without anticoagulation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fractional Flow Reserve: Patients with suspected coronary artery disease undergoing FFR to assess physiological significance of stenosis
  Interventions: Procedure: Fractional Flow Reserve

INTERVENTIONS:
Procedure: Fractional Flow Reserve — Fractional Flow Reserve performed without anticoagulation

SUMMARY:
The purpose of this study is to assess the safety of performing fractional flow reserve (FFR) of the myocardium without using anticoagulation by performing a retrospective review of 100 consecutive patients who have undergone this procedure during diagnostic catheterization.

DETAILED DESCRIPTION:
An experienced interventional cardiologist can perform FFR in a brief period of time. This procedure can safely be performed without anticoagulation, thereby lowering the associated procedural risks by avoiding the bleeding and groin complications that may occur with anticoagulation. Performing FFR without anticoagulation may also decrease facility costs as femoral artery closure can be performed using standard protocols for a diagnostic procedure, instead of standard protocols for an interventional procedure when a patient has been anticoagulated. Performing FFR without anticoagulation does not increase risk of injury to the coronary artery or thrombus in the coronary artery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate stenosis who underwent FFR without anticoagulation

Exclusion Criteria:

* Therapeutic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent fractional flow reserve (FFR) by Dr. Jonathan Roberts without anticoagulation during diagnostic catheterization were included in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Complications related to use of pressure wire | 0-30 days (index procedure)

SECONDARY OUTCOMES:
Complications due to FFR procedure | 0-30 days (index hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Roberts, MD, Principal Investigator — Clinyx, LLC